CLINICAL TRIAL: NCT01984138
Title: REVIVE: Replens Versus Intra-Vaginal Estrogen for the Treatment of Vaginal Dryness on Aromatase Inhibitor Therapy
Acronym: REVIVE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Polly A. Niravath, MD (Other)
Responsible Party: Sponsor-Investigator, Polly A. Niravath, MD, Assistant Professor, The Methodist Hospital Research Institute
Organization: The Methodist Hospital Research Institute (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: REVIVE
Record Dates: First submitted 2013-10-08; First posted 2013-11-14 (Estimated); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Estrogen Receptor Positive Breast Cancer; Breast Cancer
Keywords: estrogen receptor positive breast cancer; breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Estradiol; Replens

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Vaginal Estrogen (Experimental): vaginal estrogen with Estring or Vagifem, per the patient's preference
  Interventions: Drug: ESTRING; Drug: Vagifem
- REPLENS (Active Comparator): Replens
  Interventions: Drug: Replens

INTERVENTIONS:
Drug: ESTRING — ESTRING (estradiol vaginal ring) is a slightly opaque ring with a whitish core containing a drug reservoir of 2 mg estradiol. Estradiol, silicone polymers and barium sulfate are combined to form the ring. When placed in the vagina, ESTRING releases estradiol, approximately 7.5 mcg per 24 hours, in a consistent stable manner over 90 days. ESTRING has the following dimensions: outer diameter 55 mm; cross-sectional diameter 9 mm; core diameter 2 mm. One ESTRING should be inserted into the upper third of the vaginal vault, to be worn continuously for three months.
  Other Names: (estradiol vaginal ring)
  Arms: Vaginal Estrogen
Drug: Replens — Replens should be applied vaginally, with a supplied applicator, three times each week.
  Arms: REPLENS
Drug: Vagifem — VAGIFEM:
  Vagifem (estradiol vaginal tablet) is a small, white round, film-coated, bi-convex vaginal insert, which measures 6 mm. Each vaginal insert contains 10 mcg of estradiol, and it is administered via disposable applicator. The insert is placed vaginally using the applicator, and it will dissolve on its own while releasing estradiol into the local tissues
  Other Names: Vagifem (estradiol vaginal tablet)
  Arms: Vaginal Estrogen

SUMMARY:
This study is investigating whether breast cancer patients who experience vaginal dryness while on anti-estrogen treatment could benefit from either vaginal estrogen or from a vaginal moisturizer called Replens.

DETAILED DESCRIPTION:
To evaluate Estring versus Replens for treatment of atrophic vaginitis in breast cancer survivors on adjuvant aromatase inhibitor therapy.

PRIMARY OBJECTIVE 1. To compare improvement of atrophic vaginitis signs and symptoms between women on the vaginal estrogen ring and those on Replens vaginal cream. 1.1 Administer a questionnaire at baseline, 4 weeks, 12 weeks, and 24 weeks to all patients which will assess vaginal dryness and vaginal itching. Over six months, we expect that patients who are receiving vaginal estrogen will have more improvement in atrophic vaginitis symptoms as compared to those women on Replens.

SECONDARY OBJECTIVES 2.1 Assess compliance with aromatase inhibitor (AI) therapy in each arm to see whether vaginal estrogen therapy increases AI compliance among women who have atrophic vaginitis. Compliance will be checked by counting pills at clinic visits at 4 weeks, 12 weeks, and 24 weeks during the study treatment period, and then every 6 months for a period of 4.5 additional years, or until completion of aromatase inhibitor therapy. We expect that compliance in the vaginal estrogen arm will be superior to that of the Replens arm.

Women over the age of 18 who have been diagnosed with stage I-III ER+ breast cancer and are currently taking adjuvant AI therapy who also complain of atrophic vaginitis symptoms including vaginal dryness, vaginal itching, frequent urinary tract infections, or dyspareunia are candidates for this study. Women also must be post-menopausal as defined by any of the following: age >55 years, history of bilateral oophorectomy, amenorrhea for 1 year with intact uterus and ovaries, or serum estradiol and FSH concentrations in the post-menopausal range along with either amenorrhea for 6 months or previous hysterectomy.

ELIGIBILITY:
Inclusion Criteria:

1. be female
2. be 18 years of age or older.
3. have stage I-III ER+ breast cancer
4. be post-menopausal as defined by any of the following: age >55 years, history of bilateral oophorectomy, amenorrhea for 1 year with intact uterus and ovaries, or serum estradiol and FSH concentrations in the post-menopausal range along with either amenorrhea for 6 months or previous hysterectomy.
5. currently take adjuvant AI therapy
6. have vaginal dryness, dyspareunia, or ≥3 urinary tract infections per year since starting AI therapy
7. Patients must agree not to use any additional estrogen during the five year study period. However, use of non-estrogen containing lubricants prior to sexual intercourse, or otherwise, is allowed.

Exclusion Criteria:

1. use of any exogenous estrogen within the preceding four weeks
2. current vaginal infection.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2013-09; Primary Completion 2025-06-03 (Actual); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
What is the number of participants that show improvement of symptoms using vaginal estrogen as compared to the control. | 4.5 years
  To compare improvement of atrophic vaginitis signs and symptoms between women on the vaginal estrogen ring and those on Replens vaginal cream. 1.1 Administer a questionnaire at baseline, 4 weeks, 12 weeks, and 24 weeks to all patients which will assess vaginal dryness and vaginal itching. Over six months, we expect that patients who are receiving vaginal estrogen will have more improvement in atrophic vaginitis symptoms as compared to those women on Replens.

SECONDARY OUTCOMES:
Compliance of use of Aromatase Inhibitor to assure safety | 4.5 years
  Assess compliance with aromatase inhibitor therapy in each arm. Assess sexual health of survivors.
  Using an ultra-sensitive estrogen assay, investigate the changes in serum estrogen levels in each arm over time. Compare the change in serum estrogen level from baseline to 6 months in the Estring arm vs. Replens arm.

OTHER OUTCOMES:
EXPLORATORY OBJECTIVE | 5 years
  To evaluate breast cancer recurrence in each arm over a 5 year time period
Evaluation of vaginal dryness by vaginal pH | 6 months from baseline
  Evaluate vaginal dryness by a potentially more objective measure - vaginal pH. We will test vaginal pH at baseline and 6 months using a pH strip and will report the pH on the research record. We expect that women on vaginal estrogen will have lower pH at 6 months, compared to women on Replens.

CONTACTS AND LOCATIONS:
Overall Officials: Polly Niravath, MD, Principal Investigator — Houston Methodist Cancer Center
Locations (1):
- Houston Methodist Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No